CLINICAL TRIAL: NCT05856006
Title: Effects of Upper Trapezius Stretching With and Without Mid Lower Trapezius Strenghthening Exercises on Pain, Disability and Quality of Life in Female Desk Workers With Trapezius Myalgia
Brief Title: Effects of Upper Trapezius Stretching With and Without Mid Lower Trapezius Strengthening in Trapezius Myalgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/23/0527
Record Dates: First submitted 2023-05-04; First posted 2023-05-12 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Trapezius Myalgia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stretching Group (Active Comparator): upper trapezius stretching plus neck isometrics
  Interventions: Other: upper trapezius stretching plus neck isometrics
- Stretching plus strengthening Group (Experimental): upper trapezius stretching with mid-lower trapezius strengthening exercises plus neck isometrics
  Interventions: Other: upper trapezius stretching with mid-lower trapezius strengthening exercises plus neck isometrics

INTERVENTIONS:
Other: upper trapezius stretching plus neck isometrics — upper trapezius stretching plus neck isometrics
  Arms: Stretching Group
Other: upper trapezius stretching with mid-lower trapezius strengthening exercises plus neck isometrics — Mid-Lower Trapezius strengthening exercise includes:
  1. Latissimus pull down
  2. Prone V- raise
  3. Modified Prone Cobra
  Arms: Stretching plus strengthening Group

SUMMARY:
A Randomized controlled trial will be conducted. Non-probability convnience sampling will be used to collect the data. Sample size of 42 subjects with age group between 18 to 40 years will be taken. Data will be collected by using tools Numeric Pain Rate Scale (NPRS) for pain, Neck Disability Index (NDI) for disability and SF-36 for Quality of life. An informed consent will be taken. A total of 20 subjects will be selected by following inclusion and exclusion criteria and will equally divided in to two groups by random number generator table. Both groups will come thrice per week for a total of 4 weeks.

DETAILED DESCRIPTION:
Trapezius myalgiais the complaint of pain, stiffness, and tightness of the upper trapezius muscle. It is characterised by acute or persistent neck-shoulder pain. In today's society, due to the increased use of computers, where the neck and shoulders are maintained in static abnormal postures to look at the computer screens and become vulnerable to cause neck pain. The aim of the study is to determine effects of upper trapezius stretching with and without mid lower trapezius strengthening exercises on pain, disability and quality of life in females with work related trapezius myalgia.

A Randomized controlled trial will be conducted in physiotherapy outpatient department of Bahria International Hospital Lahore. Non-probability convnience sampling will be used to collect the data. Sample size of 42 subjects with age group between 18 to 40 years will be taken. Data will be collected by using tools Numeric Pain Rate Scale (NPRS) for pain, Neck Disability Index (NDI) for disability and SF-36 for Quality of life. An informed consent will be taken. A total of 20 subjects will be selected by following inclusion and exclusion criteria and will equally divided in to two groups by random number generator table. Both groups will come thrice per week for a total of 4 weeks. The data will be analysed using SPSS software version 25. After assessing normality of data by Shapiro-Wilk test, it will be decided either parametric or non-parametric test will be used within a group or between two groups.

ELIGIBILITY:
Inclusion Criteria:

* • Females between the age range of 18-40 years

  * Examination-Symptoms provoked by neck movement and palpation of Trapezius musculature.
  * Positive Trapezius Strength Test

Exclusion Criteria:

* Participants who present with dizziness and vertigo
* Infection or febrile state at the time of performing the test;
* Anxiety or extreme emotional tension;
* pharmacological treatment (analgesics, muscle relaxants, anxiolytics, antidepressants)
* Disc lesions

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 40 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-09-15 (Actual)

PRIMARY OUTCOMES:
Numeric Pain Rate Scale (NPRS) | up to 4 weeks
  Patient level of pain will be assessed using this scale. This scale ranges from 0to10."0"indicates "no pain" and "10" indicates "worst pain".
Neck Disability Index | up to 4 weeks
  NDI is a 10-item questionnaire that measures a patient's self-reported neck pain related disability
SF-36 for Quality of life | up to 4 weeks
  The SF-36 is a 36-item scale constructed to survey health status and quality. The SF-36 assesses eight health concepts: limitations in Quality of lifephysical activities because of health problems; limitations in social activities because of physical or emotional problems; limitations in usual role activities because of physical health problems); bodily pain; general mental health (psychological distress and well-being); limitations in usual role activities because of emotional problems; vitality (energy and fatigue); and general health perceptions. The standard form of the instruments asks for participants to reply to questions according to how they have felt over the previous week. The items use Likert-type scales, some with 5 or 6 points and others with 2 or 3 pointsmotions

CONTACTS AND LOCATIONS:
Overall Officials: Maryam Azam, MS*, Principal Investigator — Riphah International University
Locations (1):
- Bahria International Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wang YZ, Wang AN, Gao XS, Du Y, Li L, Zhao JJ. [Effect of the small needle knife through the Zusanli(ST 36) on behavior and hippocampal expression of NLRP3 and IL-1beta in myalgia comorbid depressed rats]. Zhongguo Gu Shang. 2019 Dec 25;32(12):1151-1155. doi: 10.3969/j.issn.1003-0034.2019.12.017. Chinese. PMID 31870077
- [Background] Kamper SJ, Henschke N, Hestbaek L, Dunn KM, Williams CM. Musculoskeletal pain in children and adolescents. Braz J Phys Ther. 2016 Feb 16;20(3):275-84. doi: 10.1590/bjpt-rbf.2014.0149. PMID 27437719
- [Background] Lee KW, Kim WH. Effect of thoracic manipulation and deep craniocervical flexor training on pain, mobility, strength, and disability of the neck of patients with chronic nonspecific neck pain: a randomized clinical trial. J Phys Ther Sci. 2016 Jan;28(1):175-80. doi: 10.1589/jpts.28.175. Epub 2016 Jan 30. PMID 26957752
- [Background] Rodriguez-Sanz J, Malo-Urries M, Lucha-Lopez MO, Lopez-de-Celis C, Perez-Bellmunt A, Corral-de-Toro J, Hidalgo-Garcia C. Comparison of an exercise program with and without manual therapy for patients with chronic neck pain and upper cervical rotation restriction. Randomized controlled trial. PeerJ. 2021 Nov 24;9:e12546. doi: 10.7717/peerj.12546. eCollection 2021. PMID 34900443
- [Background] Cote P, Cassidy JD, Carroll L. The Saskatchewan Health and Back Pain Survey. The prevalence of neck pain and related disability in Saskatchewan adults. Spine (Phila Pa 1976). 1998 Aug 1;23(15):1689-98. doi: 10.1097/00007632-199808010-00015. PMID 9704377
- [Background] Suvarnnato T, Puntumetakul R, Kaber D, Boucaut R, Boonphakob Y, Arayawichanon P, Chatchawan U. The effects of thoracic manipulation versus mobilization for chronic neck pain: a randomized controlled trial pilot study. J Phys Ther Sci. 2013 Jul;25(7):865-71. doi: 10.1589/jpts.25.865. Epub 2013 Aug 20. PMID 24259872
- [Background] Chansirinukor W, Wilson D, Grimmer K, Dansie B. Effects of backpacks on students: measurement of cervical and shoulder posture. Aust J Physiother. 2001;47(2):110-6. doi: 10.1016/s0004-9514(14)60302-0. PMID 11552866
- [Background] Lee KS, Lee JH. Effect of maitland mobilization in cervical and thoracic spine and therapeutic exercise on functional impairment in individuals with chronic neck pain. J Phys Ther Sci. 2017 Mar;29(3):531-535. doi: 10.1589/jpts.29.531. Epub 2017 Mar 22. PMID 28356648